CLINICAL TRIAL: NCT00597701
Title: Treating Alcohol Withdrawal With Oral Baclofen: a Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Treating Alcohol Withdrawal With Oral Baclofen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essentia Health (Other)
Responsible Party: Jeffrey Lyon, MD, Essentia Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 090403
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Results first posted 2011-07-26 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Alcohol Withdrawal Delirium
Keywords: Alcohol withdrawal; Delirium tremors
MeSH Terms: conditions — Alcohol Withdrawal Delirium | interventions — Baclofen; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baclofen (Active Comparator): Standard benzodiazepine therapy plus baclofen 10 mg every 8 hours for 72 hours (9 doses) as an inpatient, or until discharge if before 72 hours.
  Interventions: Drug: Baclofen; Drug: Lorazepam
- Placebo (Placebo Comparator): Standard benzodiazepine therapy plus placebo every eight hous as inpatients for 72 hours or until discharge if less than 72 hours.
  Interventions: Drug: Placebo; Drug: Lorazepam

INTERVENTIONS:
Drug: Baclofen — Baclofen 10 mg by mouth every 8 hours for 72 hours or until discharge if before 72 hours.
  Other Names: Lioresal
  Arms: Baclofen
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Lorazepam — Lorazepam was provided to all subjects (both arms of the study), as indicated by clinical condition. Standard "symptom-triggered dosing" of lorazepam for alcohol withdrawal was used. That is, the size and the frequency of the dose of lorazepam was determined by the severity of the alcohol withdrawal symptoms.

SUMMARY:
The purpose of this study is determine if subjects with alcohol withdrawal who receive oral baclofen, plus standard benzodiazepine therapy, will experience less severe withdrawal symptoms than those who receive placebo plus standard benzodiazepine therapy.Subjects with alcohol withdrawal syndrome(AWS)who receive baclofen plus standard benzodiazepine therapy will experience fewer complications of AWS (as measured by use of additional sedatives, restraints, and/or intensive care unit [ICU] admissions) compared with subjects who receive placebo plus standard benzodiazepine therapy.

DETAILED DESCRIPTION:
Alcohol use is ubiquitous in American society. 83% of Americans have ever consumed alcohol, 51% have in the lst month.

The average American consumes 2.18 gallons of ethanol yearly. Alcohol related morbidity and mortality are staggering problems in the USA. Symptoms of alcohol withdrawal occur because alcohol is a central nervous system depressant; abrupt withdrawal unmasks compensatory overactivity of certain parts of the nervous system, including sympathetic autonomic outflow. 5% of patients who undergo alcohol suffer from Delirium Tremors (DTs), a syndrome characterized by hallucinations, disorientation, tachycardia, hypertension, low grade fever, agitation, and diaphoresis.

DTs typically begin between 48-96 hours after the last drink and last 1 to 5 days. DTs requires hospitalization and vigorous activity in an ICU setting.

The most successful drug treatment for alcohol withdrawal has been found to be the benzodiazepines.

Symptom triggered treatment was found to be as effective as a fixed dose treatment to result in less drug being used overall, with a trend toward shorter duration of withdrawal treatment.

Baclofen is used orally for the treatment of spasticity resulting from multiple sclerosis, spinal cord injuries/diseases and intrathecally for spasticity related to cerebral palsy, spinal cord injury, and amyotrophic lateral sclerosis (ALS).

Its proposed benefit in alcohol withdrawal is that it may reduce voluntary alcohol intake, alcohol craving, and may suppress the intensity of alcohol withdrawal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual, 4th version, revised (DSMr-IV) criteria for alcohol withdrawal syndrome (AWS).
* Be an inpatient at St. Mary's Medical Center (SMMC) or Miller Dwan Medical Center (MDMC) at time of study enrollment.
* Have an alcohol withdrawal score as measured by standard SMMC or MDMC inpatient protocol sufficient to trigger the use of benzodiazepine withdrawal therapy.
* Agree to abstain for alcohol for duration of study.
* Be able to provide informed consent.

Exclusion Criteria:

* The patient must not have any other active drug dependence in addition to alcohol.
* Be unwilling or unable to forgo alcohol for the duration of the study.
* Be using baclofen at the time of study enrollment.
* Be using benzodiazepines for any reason other than acute alcohol withdrawal syndrome at time of study enrollment.
* have known baclofen or benzodiazepine sensitivity.
* Be unable to take oral (PO) meds.
* Be unable to complete one of two consenting procedures.
* Be pregnant or breastfeeding.
* Have a serum creatine level > 2.0.
* Have a history of non alcoholic withdrawal seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2003-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lyon, MD, Principal Investigator — Essentia Health
Locations (1):
- Essentia Health, Duluth, Minnesota, United States

REFERENCES:
- [Background] Colombo G, Agabio R, Carai MA, Lobina C, Pani M, Reali R, Addolorato G, Gessa GL. Ability of baclofen in reducing alcohol intake and withdrawal severity: I--Preclinical evidence. Alcohol Clin Exp Res. 2000 Jan;24(1):58-66. PMID 10656194
- [Background] Addolorato G, Caputo F, Capristo E, Janiri L, Bernardi M, Agabio R, Colombo G, Gessa GL, Gasbarrini G. Rapid suppression of alcohol withdrawal syndrome by baclofen. Am J Med. 2002 Feb 15;112(3):226-9. doi: 10.1016/s0002-9343(01)01088-9. No abstract available. PMID 11893350

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy-nine subjects met study inclusion criteria, and provided informed consent for participation in the study.
Pre-assignment Details: Of 79 enrolled subjects, 44 developed signs of Alcohol Withdrawal Syndrome (AWS) sufficient to meet Diagnostic and Statistical Manual, 4th version, revised (DSMr-IV) criteria for AWS. These 44 were randomized to receive baclofen or placebo, in addition to benzodiazepine therapy. Of the 44 subjects randomized, 31 completed 72 hours of observation.
Period: Overall Study
Arm/Group | Baclofen | Placebo
Started | 25 | 21
Completed | 18 | 13
Not Completed | 7 | 8
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Death | 0 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Did not start intervention (pharmacy er) | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baclofen | Placebo | Total
Number analyzed (Participants) | 25 | 19 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 18 | 42
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 47.5 (10.3) | 46.1 (11.9) | 46.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 19 | 18 | 37
Region of Enrollment [Number; unit: participants]
  United States | 25 | 19 | 44

OUTCOME MEASURES:

1. Primary Outcome: Benzodiazepine Doses Used to Treat Acutely-withdrawing Alcoholic Patients in the Baclofen-treated and Placebo-treated Groups
Description: In acutely-withdrawing alcoholic patients treated with either baclofen or placebo, symptom-driven benzodiazepine doses were assessed for the 72 hours following the first Clinical Institute Withdrawal Assessment (CIWA) score of 11 or greater.
Time Frame: From eligibility for randomization (Clinical Institute Withdrawal Assessment [CIWA] score of at least 11) until 72 hours of observation had been completed.
Measure: Mean (Standard Deviation); unit: mg of benzodiazepine per 8 hours
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 25 | 21
mg of benzodiazepine per 8 hours | 14.1 (8.9) | 124.4 (290.3)

ADVERSE EVENTS:
Arm/Group | Baclofen | Placebo
Serious Adverse Events (participants affected / at risk) | 2/25 | 1/19
Other Adverse Events (participants affected / at risk) | 0/25 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baclofen (N=25) | Placebo (N=19)
Rapid progression of complications of alcoholism (General disorders) | 2 (2) | 1 (1) — Alcohol withdrawal - complications

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No